CLINICAL TRIAL: NCT06919679
Title: Phase II Trial of BrECADD in HIV-Positive Patients With Advanced-Stage Classical Hodgkin Lymphoma
Acronym: BASTION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5576; 2025-521749-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma (Category)
Keywords: advanced stage; HIV positive; Brentuximab Vedotin
MeSH Terms: conditions — Hodgkin Disease; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Participants receive chemotherapy with BrECADD in standard doses and cycle length. After the first two cycles, a restaging is performed by contrast-enhanced computed tomography (ceCT) and PET (PET/CT) in order to guide response-adapted continuation of therapy consisting of 4 or only 2 additional cycles of BrECADD in case of a PET-positive or -negative staging result, respectively.
  Interventions: Drug: BrECADD

INTERVENTIONS:
Drug: BrECADD — Brentuximab Vedotin Etoposide Cyclophosphamide Doxorubicin Dacarbacine Dexamethasone

SUMMARY:
Participants receive chemotherapy with BrECADD in standard doses and cycle length. After the first two cycles, a restaging is performed by contrast-enhanced computed tomography (ceCT) and PET (PET/CT) in order to guide response-adapted continuation of therapy consisting of 4 or only 2 additional cycles of BrECADD in case of a PET-positive or -negative staging result, respectively. A second restaging will be performed after completion of chemotherapy. In patients with PET-positive residual disease, local irradiation followed by another restaging is recommended. ART should be continued during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed first diagnosis of cHL
* Advanced-stage disease: stage IIB with large mediastinal mass and/or extranodal lesions or stage III or IV
* No previous treatment for HL with the exception of steroid prephase
* Confirmed HIV infection with CD4 counts ≥ 150/μL at registration or > 250/μL at any time within 8 months prior to HL diagnosis
* Continuation of antiretroviral treatment (ART) / Initiation of ART in patients who are ART-naive
* Age: 18-60 years

Exclusion Criteria:

* Previous malignancy during last 5 years or active malignancy, prior chemotherapy or radiotherapy which precludes protocol treatment
* Nodular lymphocyte-predominant Hodgkin lymphoma or composite lymphoma
* Multi-drug resistant HIV infection or concurrent AIDS-defining conditions
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | PFS at 1 year